CLINICAL TRIAL: NCT04614077
Title: Vascular Graft Storage Solution Preserves Endothelial Function
Acronym: VGE
Status: Completed | Type: Observational
Sponsor: Klinikum Floridsdorf (Other)
Responsible Party: Principal Investigator, Bernhard Winkler, Associate Professor Priv. Doz. DDR., Associate Professor MD, Klinikum Floridsdorf
Other Study IDs: A2020
Record Dates: First submitted 2020-10-04; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Vein Injury
Keywords: vein; preservation; endothelium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A( saline): The vein piece 1 cm is taken from one patient, then the piece is divided and assigned to saline or the specific solution.
  Interventions: Other: ex vivo organ bath testing, preservation of vein sections without contact to patient
- B specific solution: The vein piece 1 cm is taken from one patient, then the piece is divided and assigned to saline or the specific solution.
  Interventions: Other: ex vivo organ bath testing, preservation of vein sections without contact to patient

INTERVENTIONS:
Other: ex vivo organ bath testing, preservation of vein sections without contact to patient — 1 piece of vein is separated during surgical bypass procedure, then randomized and put ex vivo in two solutions: saline and specific solution, then tested in the organ bath
  Other Names: organ bath ex vivo comparing saline vs specific solution

SUMMARY:
Since Saline is still the most widely used storage and flushing solution in cardiovascular procedures despite knowing evidence of its influence on the human endothelial cell function the main aim of this study was to assess the effect of DuraGraft©, an intraoperative graft treatment solution, on human saphenous vein segments 8 Remnants from the operation after trimming the bypass length), rat aortic segments and human umbilical vein endothelial cells (HUVECs) in comparison to saline.

DETAILED DESCRIPTION:
Saline is still the most widely used storage and flushing solution in cardiovascular procedures despite knowing evidence of its influence on the human endothelial cell function. Aim of this study was to assess the effect of DuraGraft©, an intraoperative graft treatment solution, on human saphenous vein segments, rat aortic segments and human umbilical vein endothelial cells (HUVECs) in comparison to saline. According to literature saline could have detrimental effects on the endothelium but data shows conflicting evidence. Duragraft a so called endothelial preservation solution should protect the human endothelium. Intent of this observational study was to study the effects of both solutions and compare them.

Within 12 patients undergoing aortocoronary bypass surgery, left overs from saphenous vein graft segments were randomized to DuraGraft© (n=12/6) or saline (n=12/6) solution before intraoperative storage. These segments as well as rat aortic segments underwent assessment of vascular function in a multichamber isometric myograph system in comparison to Krebs-Henseleit solution (KHS), a physiologic organ buffer solution. Additionally, human umbilical vein endothelial cells (HUVECs) were used for cell viability tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing isolated CABG procedure or CABG plus aortic or mitral valve surgery with at least one saphenous vein or radial artery grafts
* Patient is ≥18 years of age
* Patient (or a legally authorized representative) is willing and able to provide consent
* DuraGraft® is being used for the CABG procedure

Exclusion Criteria:

* Participation in a device study or receiving active drug product in an investigational study within one month (30 days) prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing bypass surgery exluding emergency cases
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
vessel function organ bath assessment | 3 hours
  defines significant contraction or relaxation between the two solutions, a myograph will be used, every change above 5 nM will be seen as significant.

SECONDARY OUTCOMES:
cell viability testing | 60 minutes
  shows significant difference between the two solutions, cell number of living cells will be simply counted and compared between the two solutions using a standard microscope and counting chamber

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Winkler, Associate Professor Priv. Doz. DDR., Principal Investigator — Klinikum Floridsdorf
Locations (1):
- KH North Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
only during publication or manuscript preparation data will be shared but no patients names or data.

REFERENCES:
- [Background] Santoli E, Di Mattia D, Boldorini R, Mingoli A, Tosoni A, Santoli C. University of Wisconsin solution and human saphenous vein graft preservation: preliminary anatomic report. Eur J Cardiothorac Surg. 1993;7(10):548-52. doi: 10.1016/1010-7940(93)90055-g. PMID 8267997
- [Background] Winkler B, Reineke D, Heinisch PP, Schonhoff F, Huber C, Kadner A, Englberger L, Carrel T. Graft preservation solutions in cardiovascular surgery. Interact Cardiovasc Thorac Surg. 2016 Aug;23(2):300-9. doi: 10.1093/icvts/ivw056. Epub 2016 Apr 10. PMID 27068248
- [Derived] Kiss A, Szabo PL, Dostal C, Arnold Z, Geisler D, Crailsheim I, Folkmann S, Grabenwoger M, Podesser BK, Winkler B. Specific Graft Treatment Solution Enhances Vascular Endothelial Function. Rev Cardiovasc Med. 2022 Oct 28;23(11):368. doi: 10.31083/j.rcm2311368. eCollection 2022 Nov. PMID 39076175